CLINICAL TRIAL: NCT00439764
Title: Health Education vs. Health Education Plus Physical Therapy for Low Back Pain Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kovacs Foundation (Other)
Collaborators: Consejería de Sanidad, Junta de Castilla y León (Unknown)
Responsible Party: Celia Albaladejo, Dirección General de Salud Pública y Consumo, Consejería de Sanidad, Junta de Castilla y León
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FK-JCL-14
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2008-11

CONDITIONS: Low Back Pain
Keywords: Low back pain, health education, physical therapy
MeSH Terms: conditions — Low Back Pain; Health Education

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Routine clinical practice and talk on general health
  Interventions: Behavioral: General health talk; Behavioral: Handout of The Back Book; Behavioral: Back exercise
- 2 (Active Comparator): Talk on back health and handout of The Back Book
  Interventions: Behavioral: Handout of The Back Book; Behavioral: Back exercise
- 3 (Active Comparator): Routine clinical practice, talk on back health, handout of The Back Book and back exercise
  Interventions: Behavioral: Back exercise

INTERVENTIONS:
Behavioral: General health talk — Routine clinical practice and talk on general health
  Arms: 1
Behavioral: Handout of The Back Book — Talk on health of the back and handout of The Back Book
  Arms: 1; 2
Behavioral: Back exercise — Routine clinical practice, talk on back health, handout of The Back Book and back exercise

SUMMARY:
The primary purpose of this study is to assess the effectiveness of a brief educational program and of an additional program in physical therapy, for the treatment of low back pain in Primary Care of the Spanish National Health Service. This is a controlled, cluster randomized community trial.

ELIGIBILITY:
Inclusion Criteria:

* Consultation for low back pain, with or without referred or radiated pain; no signs of systemic disease or criteria for surgery.

Exclusion Criteria:

* Inability to fill out the questionnaires (blindness, dementia, illiteracy; total habitual prostration;
* Diagnosis of rheumatologic inflammatory disease, fibromyalgia or cancer in last 5 years;
* Suspicion of fibromyalgia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Intensity of pain, measured at baseline, 90, and 180 days later | 6 months
Disability, measured at baseline, 90, and 180 days later | 6 months
Sick leave, measured at baseline, 90, and 180 days later | 6 months

SECONDARY OUTCOMES:
Fear avoidance beliefs, measured at baseline, 90, and 180 days later | 6 months
Quality of life, measured at baseline, 90, and 180 days later | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Chair — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Celia Albaladejo, MD, Study Director — Consejería de Sanidad, 47071 Valladolid, Spain; Rafael del Pino, PT, Principal Investigator — Centro de Especialidades de Fisioterapia, 47014 Valladolid, Spain
Locations (1):
- Servicio de Atención Primaria del SACYL, Valladolid, Castille and León, Spain

REFERENCES:
- [Background] Burton AK, Waddell G, Tillotson KM, Summerton N. Information and advice to patients with back pain can have a positive effect. A randomized controlled trial of a novel educational booklet in primary care. Spine (Phila Pa 1976). 1999 Dec 1;24(23):2484-91. doi: 10.1097/00007632-199912010-00010. PMID 10626311
- [Background] Cherkin DC, Eisenberg D, Sherman KJ, Barlow W, Kaptchuk TJ, Street J, Deyo RA. Randomized trial comparing traditional Chinese medical acupuncture, therapeutic massage, and self-care education for chronic low back pain. Arch Intern Med. 2001 Apr 23;161(8):1081-8. doi: 10.1001/archinte.161.8.1081. PMID 11322842
- [Background] Frost H, Lamb SE, Doll HA, Carver PT, Stewart-Brown S. Randomised controlled trial of physiotherapy compared with advice for low back pain. BMJ. 2004 Sep 25;329(7468):708. doi: 10.1136/bmj.38216.868808.7C. Epub 2004 Sep 17. PMID 15377573
- [Derived] Albaladejo C, Kovacs FM, Royuela A, del Pino R, Zamora J; Spanish Back Pain Research Network. The efficacy of a short education program and a short physiotherapy program for treating low back pain in primary care: a cluster randomized trial. Spine (Phila Pa 1976). 2010 Mar 1;35(5):483-96. doi: 10.1097/BRS.0b013e3181b9c9a7. PMID 20147875
- See also: Spanish Back Pain Research Network site that describes objectives and projects of its members. — http://www.reide.org